CLINICAL TRIAL: NCT03484000
Title: The ONE-MIND Study: Evaluating the Efficacy of Online Mindfulness-Based Cancer Recovery (MBCR) During Chemotherapy Treatment (CT) to Impact Fatigue, Side Effects and Quality of Life (QL) in a Randomized Waitlist Controlled Trial
Brief Title: The ONE-MIND Study: Evaluating the Efficacy of Online Mindfulness-Based Cancer Recovery During Chemotherapy Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Linda E. Carlson, Enbridge Research Chair in Psychosocial Oncology, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HREBA.CC-18-0028
Record Dates: First submitted 2018-03-24; First posted 2018-03-30 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer; Colorectal Cancer; Chemotherapy Effect
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate MBCR group (Experimental): The Online Mindfulness Based Cancer Recovery (MBCR) program intervention is delivered in 12 weekly real-time interactive 55-minute sessions offered over consecutive weeks.
  Interventions: Behavioral: Online Mindfulness Based Cancer Recovery (MBCR)
- Waitlist control group (Other): Treatment as usual, followed by a delayed (wait-list) intervention of the same Online Mindfulness Based Cancer Recovery (MBCR) program after the post-CT assessment.
  Interventions: Behavioral: Online Mindfulness Based Cancer Recovery (MBCR)

INTERVENTIONS:
Behavioral: Online Mindfulness Based Cancer Recovery (MBCR) — MBCR is a group behavioral treatment that trains participants in mindfulness techniques through meditation and gentle mindful movement

SUMMARY:
Background: Chemotherapy treatment (CT) can have burdensome side effects such as fatigue, nausea-vomiting, and sleep problems that can significantly affect patients' quality of life. Fatigue is the most common, lasting and bothersome of these, which prevents people from working and carrying out daily activities. Mindfulness-Based Cancer Recovery (MBCR) is an evidence-based group training program which has shown to help treat negative physical and psychosocial symptoms in cancer patients. The investigators propose to evaluate a pilot-tested online-MBCR program for patients undergoing CT who may be low on energy, time or have compromised immunity.

Objectives: To evaluate the impact of participation in online MBCR during CT on fatigue (primary outcome), sleep, pain, nausea/vomiting, mood disturbance, stress symptoms and quality of life (secondary outcomes) as well as cognitive function and return to work (exploratory outcomes) over the course of treatment.

Methods: The study design is a randomized wait-list controlled trial, conducted during CT for patients with breast or colorectal cancer. Participants will take the 12-week online MBCR program at home within 2 weeks of randomization (immediate group) or after CT completion (waitlist group). Outcomes will be assessed online at, 1) Baseline, 2) Post-MBCR, 3) Post-CT (primary outcome) and 4) 12 months post-baseline.

Anticipated Findings: MBCR is a promising adjuvant program that could help patients prevent, delay or diminish aversive symptoms and side-effects associated with CT, particularly fatigue. If helpful, online-MBCR could be made easily available at cancer centers worldwide and significantly lessen the burden of cancer treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women over the age of 18
2. Diagnosed with either a) stage I-III HER 2 normal breast carcinoma or b) Stage II-III colorectal carcinoma
3. Scheduled to undergo either neoadjuvant or adjuvant: a) FEC- D or AC-T chemotherapy or b) FOLFOX or CAPEOX chemotherapy
4. Weekly access to high-speed internet
5. Access to a computer/tablet/smart phone
6. Able to attend MBCR classes at scheduled times
7. Sufficient ability to speak and read English
8. Willingness to be randomized into immediate or waitlist groups and complete all assessments

Exclusion Criteria:

1. Metastatic patients
2. Suffering from current Major Depressive Disorder, Bipolar Disorder or other psychiatric disorder (self-report)
3. Currently engaging in meditation one or more times per week within the previous year.
4. Participation in an MBCR or MBSR program in the last five years.
5. Cognitive impairment (>6 on the Brief Screen for Cognitive Impairment)
6. Physical functional impairment that would interfere with the ability to participate in the intervention (on the PAR-Q questionnaire)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Fatigue | 6 months
  Fatigue will be measured by the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F 68) is the most commonly-used cancer-related fatigue scale. Using a 5-point Likert scale (from "not at all" to "very much"), the 13-items reflect participants' specific fatigue concerns in the past 7 days. The total score has well-established norms both in the literature and from our prior work and shows responsiveness to intervention

CONTACTS AND LOCATIONS:
Overall Officials: Linda E Carlson, PhD, Principal Investigator — University of Calgary; Barry D Bultz, PhD, Study Chair — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Subnis UB, Farb NA, Piedalue KL, Speca M, Lupichuk S, Tang PA, Faris P, Thoburn M, Saab BJ, Carlson LE. A Smartphone App-Based Mindfulness Intervention for Cancer Survivors: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 May 11;9(5):e15178. doi: 10.2196/15178. PMID 32390591